CLINICAL TRIAL: NCT01053156
Title: Randomized Double-Blind Controlled Cross Over Trial of Minocycline in Children With Fragile X Syndrome
Brief Title: Trial of Minocycline to Treat Children With Fragile X Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: The National Fragile X Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 200917522
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Results first posted 2014-07-30 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X syndrome; minocycline; targeted treatment
MeSH Terms: conditions — Fragile X Syndrome; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo pill (Placebo Comparator): All patients will be on placebo for 3 months in this crossover study.
  Interventions: Drug: Placebo
- Minocycline (Experimental): All patients will be on minocycline for 3 months in this crossover trial.
  Interventions: Drug: minocycline hydrochloride

INTERVENTIONS:
Drug: minocycline hydrochloride — Minocycline hydrochloride dosed orally once a day for 3 months.
  Arms: Minocycline
Drug: Placebo — Placebo will be given daily for 3 months.
  Arms: Placebo pill

SUMMARY:
This is a single center study at the UC Davis MIND Institute in patients age 3.5-16 years of age with fragile X syndrome (FXS), funded by a National Fragile X Foundation Grant. It is a controlled trial of minocycline, an antibiotic commonly used in children for infection or for treatment of neurodegenerative disorders. We are investigating its use in FXS because it lowers matrix metalloproteinase 9 (MMP9) levels, which are high in FXS, and it also strengthens brain connections in the animal models of FXS. We hypothesize that minocycline will likely be helpful for language, behavior and/or cognition in fragile X patients.

DETAILED DESCRIPTION:
This is a single center study at the UC Davis MIND Institute in patients age 3.5-16 years of age with fragile X syndrome (FXS), funded by a National Fragile X Foundation Grant. It is a controlled trial of minocycline, an antibiotic commonly used in children for infection or for treatment of neurodegenerative disorders. We are investigating its use in FXS because it lowers matrix metalloproteinase 9 (MMP9) levels, which are high in FXS, and it also strengthens brain connections in the animal models of FXS. We hypothesize that minocycline will likely be helpful for language, behavior and/or cognition in fragile X patients.

The aim of this study is to carry out a double-blind placebo controlled trial of minocycline treatment in children with FXS who are 3.5 to 16 years of age. At baseline, we will assess behavior and perceptual and cognitive development. After the children have been treated for 3 months with either minocycline or placebo, they undergo the same baseline testing. They will then cross over and be treated for a second 3 months. We will carry out testing again at the end of the second 3 month period. We will also assess the side effects of minocycline treatment throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Must have fragile X syndrome with molecular documentation
* Current pharmacological treatment regimen has been stable for at least 4 weeks

Exclusion Criteria:

* Subjects who plan to initiate or change pharmacologic or non-pharmacologic interventions during the course of the study
* subjects who are unable to take oral medication
* subjects who have been on minocycline previously
* subjects who are allergic to minocycline or tetracyclines
* subjects who are pregnant
* subjects with history of lupus or hepatic dysfunction

Ages: 42 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randi J Hagerman, MD, Principal Investigator — M.I.N.D. Institute at University of California at Davis, Sacramento CA
Locations (1):
- M.I.N.D. Institute at University of California at Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Background] Bilousova TV, Dansie L, Ngo M, Aye J, Charles JR, Ethell DW, Ethell IM. Minocycline promotes dendritic spine maturation and improves behavioural performance in the fragile X mouse model. J Med Genet. 2009 Feb;46(2):94-102. doi: 10.1136/jmg.2008.061796. Epub 2008 Oct 3. PMID 18835858

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from January 2010 to June 2011, with the last participants completing the study in December 2011. The study site was a single site, the MIND Institute at the University of California Davis Medical Center.
Pre-assignment Details: Inclusion criteria: FXS confirmed by FMR1 DNA, age 3.5-16 years and stable pharmacological regimen > 4 weeks prior to study. Exclusion criteria:previous minocycline treatment, plans to change pharmacological intervention or allergy to tetracyclines. 66 patients enrolled; 55 patients with any data on outcome measures analyzed (11 withdrawn).
Groups:
- Minocycline First, Then Placebo Second: Minocycline hydrochloride dosed orally once a day for 3 months, the switched to placebo dosed orally once a day for 3 months.
- Placebo First, Minocycline Second: Placebo will be given once daily for 3 months, then minocycline dosed once daily for 3 months
Period: First Intervention (Week 1-12)
Arm/Group | Minocycline First, Then Placebo Second | Placebo First, Minocycline Second
Started | 33 | 33
Completed | 28 | 27
Not Completed | 5 | 6
Period: Second Intervention (Week 13-24)
Arm/Group | Minocycline First, Then Placebo Second | Placebo First, Minocycline Second
Started | 28 | 27
Completed | 26 | 22
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Population: The baseline participants are different in number from those started in the participant flow module because in our intent to treat analysis, only those who completed one or more treatment periods were included in the analysis.
Groups:
- Minocycline First, Placebo Second: Minocycline hydrochloride dosed orally once a day for 3 months, the switched to placebo dosed orally once a day for 3 months.
- Total: Total of all reporting groups
Arm/Group | Minocycline First, Placebo Second | Placebo First, Minocycline Second | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 27 | 55
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.01 (3.76) | 9.4 (3.39) | 9.21 (3.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 23 | 24 | 47
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression Scale (CGI)
Description: The CGI-I utilizes history from primary caregivers and incorporates it into a seven step clinical rating for follow up throughout treatment, from 1 "very much improved" to 7 "very much worse". Lower scores indicate more improvement. Scores were obtained post treatments. Scores from when the patients were on minocycline either first or second were combined and averaged to determine a least squares mean and placebo scores were obtained in the same manner.
Time Frame: 3 months (post first treatment) and 6 months (post second treatment)
Population: Any participant who completed at least the first arm of the trial were included in the intention to treat analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Minocycline: Minocycline dosage was assigned based on weight, with patients weighing up to 25 kg receiving 25mg once daily, those weighing between 25 and 45 kg receiving 50 mg once daily, and those weighing >45 kg receiving 100 mg once daily.
- Placebo: Placebo dosage was assigned based on weight, with patients weighing up to 25 kg receiving 25mg once daily, those weighing between 25 and 45 kg receiving 50 mg once daily, and those weighing >45 kg receiving 100 mg once daily.
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 55 | 55
units on a scale | 2.49 (0.13) | 2.97 (0.13)

2. Primary Outcome: Visual Analogue Scale- Behavior 1
Description: A VAS is used to represent a caregiver's assessment of given behaviors, which were chosen by the parents. Caregivers marked a 10 cm horizontal line representing a visual continuum of each behavior from "worst behavior" to "behavior not a problem." Greater values indicate greater improvement. This measure represents the first behavior that the caregivers noted, out of three.
Time Frame: Baseline, 3 months, 6 months
Population: Any participant who completed at least the first arm of the trial were included in the intention to treat analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Baseline: Prior to any intervention being started.
Arm/Group | Baseline | Minocycline | Placebo
Number analyzed (Participants) | 55 | 55 | 55
units on a scale | 2.28 (0.21) | 4.60 (0.31) | 4.44 (0.30)

3. Secondary Outcome: Visual Analogue Scale- Behaviors 2
Description: A VAS is used to represent a caregiver's assessment of given behaviors, which were chosen by the parents. Caregivers marked a 10 cm horizontal line representing a visual continuum of each behavior from "worst behavior" to "behavior not a problem." Greater values indicate greater improvement. This measure represents the second behavior that the caregivers noted, out of three.
Time Frame: Baseline, 3 months, 6 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Minocycline | Placebo
Number analyzed (Participants) | 55 | 55 | 55
units on a scale | 2.62 (0.23) | 4.91 (0.31) | 4.16 (0.29)

4. Secondary Outcome: Expressive Vocabulary Test-2
Description: The EVT-2 standard score assesses language development through a participant's one word synonym response to visual stimuli. Standard scores range from 20-160. A standard score of 100 is average, with a 15 point standard deviation. Higher values represent a better outcome.
Time Frame: Baseline, 3 months and 6 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Minocycline | Placebo
Number analyzed (Participants) | 55 | 55 | 55
units on a scale | 65.92 (3.61) | 68.86 (1.28) | 67.91 (1.20)

5. Secondary Outcome: Vineland Adaptive Behavior Scale-II (VABS-II)Adaptive Behavior Composite Score
Description: The VABS-II Adaptive Behavior Composite Score was used to assess adaptive skills. An Adaptive Behavior Composite Score may range from 20-160 with an average of 100 with a standard deviation of 15. Higher scores show improvement.
Time Frame: Baseline, 3 months, and 6 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Minocycline | Placebo
Number analyzed (Participants) | 55 | 55 | 55
units on a scale | 69.88 (2.00) | 70.85 (0.92) | 71.43 (0.90)

6. Secondary Outcome: Aberrant Behavior Checklist-Community Edition (ABC-C)Composite Score
Description: The ABC-C composite scores were used to quantify the severity of a patient's behaviors. A composite score consists of subscale scores including Irritability and Agitation, Lethargy and Social Withdrawal, Stereotypic Behavior, Hyperactivity and Noncompliance, and Inappropriate Speech. The composite score may range from 0-174. Lower scores indicate improvement.
Time Frame: Baseline, 3 months, and 6 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Minocycline | Placebo
Number analyzed (Participants) | 55 | 55 | 55
units on a scale | 41.22 (3.44) | 44.22 (3.02) | 41.81 (2.94)

7. Secondary Outcome: Visual Analogue Scale Behavior 3- VAS3
Description: A VAS is used to represent a caregiver's assessment of given behaviors, which were chosen by the parents. Caregivers marked a 10 cm horizontal line representing a visual continuum of each behavior from "worst behavior" to "behavior not a problem." Greater values indicate greater improvement. This measure represents the third behavior that caregivers noted, out of three.
Time Frame: Baseline, 3 months, 6 months
Population: This behavior was not provided by all of the participating caregivers, and so the number is less than the participants analyzed for other measures.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Minocycline | Placebo
Number analyzed (Participants) | 50 | 50 | 50
units on a scale | 2.80 (0.27) | 4.88 (0.36) | 4.13 (0.35)

8. Secondary Outcome: VAS Categorized by Behavior: Aggression/ ADHD
Description: A VAS is used to represent a caregiver's assessment of given behaviors, which were chosen by the parents. Caregivers marked a 10 cm horizontal line representing a visual continuum of each behavior from "worst behavior" to "behavior not a problem." Greater values indicate greater improvement. This measure represents the least squares mean of all behaviors having to do with aggression or ADHD behaviors.
Time Frame: Baseline, 3 months, 6 months
Population: In this ad hoc analysis, the various behaviors captured on the VAS were categorized and any behaviors regarding ADHD or Aggression symptoms were placed into this category. As not every caregiver named a behavior related to ADHD or aggression, this number is less than the number of participants.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Minocycline | Placebo
Number analyzed (Participants) | 46 | 46 | 46
units on a scale | 2.38 (0.20) | 4.49 (0.32) | 4.26 (0.32)

9. Secondary Outcome: VAS Categorized by Behavior:Anxiety/ Mood
Description: A VAS is used to represent a caregiver's assessment of given behaviors, which were chosen by the parents. Caregivers marked a 10 cm horizontal line representing a visual continuum of each behavior from "worst behavior" to "behavior not a problem." Greater values indicate greater improvement. This measure represents the least squares mean of all behaviors having to do with anxiety or mood related behaviors.
Time Frame: Baseline, 3 months, 6 months
Population: In this ad hoc analysis, the various behaviors captured on the VAS were categorized and any behaviors regarding anxiety or mood symptoms were placed into this category. As not every caregiver named a behavior related to anxiety or mood, this number is less than the number of participants.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Minocycline | Placebo
Number analyzed (Participants) | 26 | 26 | 26
units on a scale | 2.47 (0.25) | 5.26 (0.46) | 4.05 (0.46)

10. Secondary Outcome: VAS Categorized by Behavior:Language/ Cognition
Description: A VAS is used to represent a caregiver's assessment of given behaviors, which were chosen by the parents. Caregivers marked a 10 cm horizontal line representing a visual continuum of each behavior from "worst behavior" to "behavior not a problem." Greater values indicate greater improvement. This measure represents the least squares mean of all behaviors having to do with language or cognitive symptoms.
Time Frame: Baseline, 3 months, 6 months
Population: In this ad hoc analysis, the various behaviors captured on the VAS were categorized and any behaviors regarding language or cognition symptoms were placed into this category. As not every caregiver named a behavior related to language or cognition, this number is less than the number of participants.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Minocycline | Placebo
Number analyzed (Participants) | 37 | 37 | 37
units on a scale | 2.58 (0.30) | 4.99 (0.37) | 4.67 (0.34)

11. Secondary Outcome: VAS Categorized by Behavior: Other
Description: A VAS is used to represent a caregiver's assessment of given behaviors, which were chosen by the parents. Caregivers marked a 10 cm horizontal line representing a visual continuum of each behavior from "worst behavior" to "behavior not a problem." Greater values indicate greater improvement. This measure represents the least squares mean of all behaviors having to do with other behaviors that were not able to be categorized.
Time Frame: Baseline, 3 months, 6 months
Population: In this ad hoc analysis, the various behaviors captured on the VAS were categorized and any behaviors not falling into the other categories were placed into this category. As not every caregiver named a behavior unrelated to the other categories, this number is less than the number of participants.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Minocycline | Placebo
Number analyzed (Participants) | 12 | 12 | 12
units on a scale | 3.49 (0.66) | 5.84 (0.54) | 3.41 (0.54)

ADVERSE EVENTS:
Arm/Group | Minocycline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/66 | 1/66
Other Adverse Events (participants affected / at risk) | 53/66 | 53/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=66) | Placebo (N=66)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) — The patient was on placebo when this occurred
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=66) | Placebo (N=66)
Diarrhea (Gastrointestinal disorders) | 15 (15) | 15 (15)
GI Upset/ Vomiting/Loss of Appetite (Gastrointestinal disorders) | 9 (9) | 15 (15)
Skin Rash/ Itching/ Swelling (Skin and subcutaneous tissue disorders) | 12 (12) | 7 (7)
Fever/Chills/URI/Sore Throat (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (11)
Headache (Nervous system disorders) | 4 (4) | 5 (5)
Sunburn/Sun Sensitivity (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Increased agitation, aggression, tantrums, uncooperative, irritability (Psychiatric disorders) | 1 (1) | 4 (4)
Blue-grey/Grey hue to teeth or other tissues (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Results may be potentially biased by study design weaknesses, including unblinding of subjects when they completed the study, drug-related side effects unblinding and preliminary efficacy analysis results known to investigators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No